CLINICAL TRIAL: NCT01868633
Title: The Effect of a Single Intraoperative Dose of Dexamethasone in Combination With Intrathecal Morphine for Post Cesarean Delivery Analgesia
Brief Title: Dexamethasone for Post Cesarean Delivery Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Unyime Ituk, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 201210765
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Pain
Keywords: Cesarean delivery; Analgesia; Pain; Dexamethasone; intrathecal morphine; spinal anesthesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Pain | interventions — Dexamethasone; Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone & spinal morphine (Active Comparator): intrathecal morphine administered at time of spinal anesthesia. After cesarean delivery 8mg (2ml) of Dexamethasone given intraoperatively
  Interventions: Drug: Dexamethasone
- Placebo injection and spinal morphine (Placebo Comparator): intrathecal morphine administered at time of spinal anesthesia. After cesarean delivery 2ml of placebo (Normal saline) drawn to mimic active drug given intraoperatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone
  Other Names: Decadron
  Arms: Dexamethasone & spinal morphine
Drug: Placebo
  Other Names: Normal saline
  Arms: Placebo injection and spinal morphine

SUMMARY:
The purpose of this study is to assess the effectiveness intravenous (IV) dexamethasone when used as part of a multimodal regimen to manage post cesarean delivery pain.

We hypothesize that a single dose of IV dexamethasone administered, as part of a multimodal analgesia after spinal anesthesia will significantly reduce post cesarean delivery opioid consumption and pain

DETAILED DESCRIPTION:
After the subjects consent to participate in the study they will be transferred to the operating room for their scheduled cesarean delivery. They will have their routine spinal anesthesia with the dosages of drugs used standardized, and a standardized regimen to manage hypotension. After delivery of the baby the subjects will be administered either the study drug or placebo depending on the randomization. The subjects will then be prescribed a standard post-operative analgesia regimen. The subjects will then be interviewed at 12,24 and 48 hours post cesarean delivery. During the interview the subjects will be asked to rate their pain, nausea and vomiting and pruritus. They will also be asked to rate their quality of recovery from the surgery using Quality of Recovery-40 questionnaire. The subjects will be contacted 6 months after the study to rate their pain using a Short-Form McGill Pain Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Non-laboring women
* Scheduled Elective Cesarean section under spinal anesthesia
* American Society of Anesthesiologists I-II physical status

Exclusion Criteria:

* Contraindications to spinal anesthesia
* allergy to study medication
* patients with allergy to morphine
* patients with uncontrolled hypertension
* history of peptic ulcer disease
* liver cirrhosis
* diabetes mellitus
* glaucoma
* known IV drug abusers
* patients with chronic pain or on long term opioids
* patients administered steroids in the past week
* women with fetuses having known congenital abnormalities
* psychiatric illness such that they are unable to comprehend or participate in study questions
* patients on antiviral medications or live virus vaccines would also be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Unyime Ituk, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Fujii Y, Nakayama M. Dexamethasone for reduction of nausea, vomiting and analgesic use after gynecological laparoscopic surgery. Int J Gynaecol Obstet. 2008 Jan;100(1):27-30. doi: 10.1016/j.ijgo.2007.07.017. Epub 2007 Sep 27. PMID 17900579 (Retraction: PMID 23599954 Int J Gynaecol Obstet. 2013 Apr;121(1):97)
- [Background] Murphy GS, Szokol JW, Greenberg SB, Avram MJ, Vender JS, Nisman M, Vaughn J. Preoperative dexamethasone enhances quality of recovery after laparoscopic cholecystectomy: effect on in-hospital and postdischarge recovery outcomes. Anesthesiology. 2011 Apr;114(4):882-90. doi: 10.1097/ALN.0b013e3181ec642e. PMID 21297442

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone & Spinal Morphine: intrathecal morphine administered at time of spinal anesthesia. After cesarean delivery 8mg (2ml) of Dexamethasone given intraoperatively
  Dexamethasone
- Placebo Injection and Spinal Morphine: intrathecal morphine administered at time of spinal anesthesia. After cesarean delivery 2ml of placebo (Normal saline) drawn to mimic active drug given intraoperatively
  Placebo
Period: Overall Study
Arm/Group | Dexamethasone & Spinal Morphine | Placebo Injection and Spinal Morphine
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone & Spinal Morphine | Placebo Injection and Spinal Morphine | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.69 (4.02) | 31.65 (5.83) | 31.67 (4.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Analgesia
Description: Comparison of postoperative opioid analgesia use between the 2 groups
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: milligrams of morphine
Arm/Group | Dexamethasone & Spinal Morphine | Placebo Injection and Spinal Morphine
Number analyzed (Participants) | 26 | 26
milligrams of morphine | 11.8 [5 to 20] | 15 [5 to 22.5]
Statistical Analysis 1: Comparison: Dexamethasone & Spinal Morphine; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Postoperative Pain at Rest and With Movement 24 Hours After Cesarean Delivery
Description: Pain scores were assessed at 6, 12 and 24 hours after surgery using a numerical rating scale (10 cm line marked at 1 cm intervals anchored on the left with "no pain" = 0 and "the worst possible pain = 10). Pain was assessed at rest and with movement
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexamethasone & Spinal Morphine | Placebo Injection and Spinal Morphine
Number analyzed (Participants) | 26 | 26
units on a scale
  Pain at rest @ 0-6hr | 1 [0 to 2] | 1 [1 to 3]
  Pain with movement @ 0-6hr | 4 [1 to 5] | 4.5 [3 to 5]
  Pain at rest @ 6-12hr | 1 [0 to 1] | 2 [1 to 3]
  Pain with movement @ 6-12hr | 3 [2 to 4] | 4 [4 to 5]
  Pain at rest @ 12-24hr | 1 [0 to 2] | 1 [1 to 3]
  Pain with movement @ 12-24hr | 4 [3 to 5] | 4 [3 to 5]

3. Secondary Outcome: Quality of Recovery
Description: Comparison of the quality of Recovery between the 2 groups using a Quality of recovery questionnaire (QoR-40). It incorporates five dimensions of health: patient support, comfort, emotions, physical independence, and pain; each item is graded on a five-point Likert scale. QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery). The scores on all 40 items are summed and the mean scores and standard deviation calculated for each study group
Time Frame: 48 hours
Population: Two patients in the dexamethasone group and 8 patients in the placebo did not complete the quality of recovery questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone & Spinal Morphine | Placebo Injection and Spinal Morphine
Number analyzed (Participants) | 24 | 18
units on a scale | 180 (10) | 177 (10)

4. Secondary Outcome: Incidence and Severity of Nausea and Pruritus
Description: Patients were asked to rate the severity of postoperative nausea using an 11-point numerical rating scale (NRS) from 0 to 10, (0: no nausea, 10: worst nausea possible). The number of vomiting episodes, if any during the 24-hour study period, was documented. Pruritus was also assessed using an 11-point NRS (0 no pruritus,10 worst pruritus possible)
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexamethasone & Spinal Morphine | Placebo Injection and Spinal Morphine
Number analyzed (Participants) | 26 | 26
units on a scale
  Nausea @ 0-6hr | 6 [2 to 10] | 2.5 [0 to 7]
  Pruritus@ 0-6hr | 5 [2 to 8] | 3 [1 to 6]
  Nausea @ 6-12hr | 0 [0 to 3] | 0 [0 to 2]
  Pruritus @ 6-12hr | 3 [2 to 7] | 0 [0 to 2]
  Nausea @12-24hr | 0 [0 to 0] | 0 [0 to 0]
  Pruritus @ 12-24hr | 2 [1 to 4] | 1 [0 to 3]

5. Other Pre Specified Outcome: Number of Participants With Chronic Pain After Cesarean Delivery
Description: Comparison of incidence of chronic pain associated with cesarean delivery between the 2 groups
Time Frame: 6 months
Population: Study participants had a telephone call follow-up 6 months after cesarean delivery by a research nurse. They were asked questions about current pain symptoms and if it is related to their cesarean delivery. Seven patients in the dexamethasone group and eight patients in the placebo did not respond when contacted
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone & Spinal Morphine | Placebo Injection and Spinal Morphine
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: A safety analysis of adverse events was done by a clinician investigator not involved in study after enrollment of every 20 patients and at the 6th-week postnatal outpatient visit( That is 6 weeks after exposure to the intervention). Adverse event data collected included surgical wound examination findings (signs of infection, poor healing, wound breakdown), postpartum blood loss and vital signs ( blood pressure, heart rate and temperature)
Arm/Group | Dexamethasone & Spinal Morphine | Placebo Injection and Spinal Morphine
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes